CLINICAL TRIAL: NCT01397201
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Parallel-group Study to Assess and Compare Efficacy and Safety of an 8-week Treatment With BI 54903 at Doses of 45.5, 90.9 and 181.8 mcg b.i.d. Administered Via Respimat® Inhaler and Fluticasone Propionate HFA 220 mcg b.i.d. in Patients With Asthma Inadequately Controlled on Low Dose ICS Therapy
Brief Title: Study on BI 54903 (Inhaled Corticosteroid) Administered Twice Daily Via Respimat Inhaler in Patients With Asthma Inadequately Controlled on Low Dose Inhaled Corticosteroid (ICS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1248.6; 2010-023168-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Results first posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

ARMS (5):
- BI 54903 - low dose (Experimental): Respimat inhaler containing low dose BI 54903 plus placebo matching hydrofluoralkane (HFA) metered dose inhaler (MDI)
  Interventions: Drug: Placebo; Drug: BI 54903
- BI 54903 - medium dose (Experimental): Respimat inhaler containing medium dose BI 54903 plus placebo matching HFA MDI
  Interventions: Drug: Placebo; Drug: BI 54903
- BI 54903 - high dose (Experimental): Respimat inhaler containing high dose BI 54903 plus placebo matching HFA MDI
  Interventions: Drug: Placebo; Drug: BI 54903
- Fluticasone propionate (Active Comparator): Fluticasone HFA MDI containing ICS plus placebo matching Respimat inhaler
  Interventions: Drug: Fluticasone propionate
- Placebo (Placebo Comparator): Placebo matching Respimat inhaler plus placebo matching HFA MDI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo matching fluticasone propionate HFA MDI
  Arms: BI 54903 - high dose; BI 54903 - low dose; BI 54903 - medium dose; Placebo
Drug: BI 54903 — BI 54903
  Arms: BI 54903 - high dose; BI 54903 - low dose; BI 54903 - medium dose
Drug: Fluticasone propionate — Fluticasone propionate
  Arms: Fluticasone propionate

SUMMARY:
The aim of the study is to assess and compare efficacy and safety of BI 54903 at 3 doses twice daily (b.i.d.), fluticasone propionate hydrofluoroalkane metered dose inhaler (HFA MDI) at a dose of 220 mcg b.i.d. and placebo b.i.d. over an 8-week treatment period in asthmatic patients aged 12 to 65 years inadequately controlled on low dose Inhaled corticosteroid (ICS) as demonstrated by a decrease in forced expiratory volume in one second (FEV1 (range 10-25%) and an asthma control questionnaire (ACQ-6) greater or equal 1.5 at time of randomisation

ELIGIBILITY:
Inclusion criteria:

1. Must be willing and able to give informed consent
2. Male and female patients aged at least 12 to 65 years
3. All patients must have a history of asthma diagnosed by a physician for at least three months at the time of enrolment into the trial according to the 2009 Global Initiative for Asthma (GINA) Guidelines. The initial diagnosis of asthma must have been made before the age of 40 years
4. All patients must be on a maintenance treatment with either medium-dose inhaled corticosteroid (ICS) plus long acting beta agonist (LABA) or high-dose inhaled corticosteroid (ICS) without long acting beta agonist (LABA), stable for at least six weeks prior to Visit 1
5. All patients must have a pre-bronchodilator forced expiratory volume in one second (FEV1) of not less than 60 to 90% of predicted normal and an asthma control questionnaire (ACQ-6) mean score of less than 1.5 at the pre-screening Visit 1
6. All patients must have an improvement in FEV1 not less than 12 % above baseline and an absolute change of at least 200 mL within 15-30 min after administration of 400 mcg salbutamol/albuterol hydrofluoroalkane metered dose inhaler (HFA MDI)
7. Patients must be never-smokers or ex-smokers with a smoking history of less than 10 pack-years and smoking cessation at least one year prior to screening
8. Patients must be able to use Respimat® inhaler and metered dose inhaler (MDI) correctly
9. Patients must be able to perform all trial-related procedures including technically acceptable pulmonary function tests and electronic peak expiratory flow (PEF) measurements, and must be able to maintain records during the study period as required in the protocol
10. To enter treatment period following additional criteria have to be met (at randomisation visit):

    * During the run-in period (at the same clinic visit) all patients must be both symptomatic (ACQ-6 mean score equal to or greater than 1.5) and have shown a decrease in morning pre-bronchodilator FEV1 not less than 10% and less than or equal to 25% from pre-screening baseline FEV1 at Visit 2.

Exclusion criteria:

1. Patients with significant pulmonary disease other than asthma or other significant medical conditions (as determined by medical history, examination and clinical investigations at screening)
2. Patients with a clinically relevant, abnormal screening haematology and/or blood chemistry finding
3. Patients with a history of upper or lower respiratory tract infection in the past four weeks prior to the pre-screening Visit 1, and during pre-screening and run-in periods
4. Patients with any exacerbation of their underlying asthma during the eight weeks prior to the pre-screening Visit 1
5. Patients with active allergic rhinitis requiring treatment with systemic corticosteroids
6. Any of the following criteria are met during the pre-screening / run-in period (Visits 1 - 6):

   * in clinic pre-bronchodilator forced expiratory volume in one second (FEV1 %) predicted less than 40%,
   * more than 12 puffs rescue salbutamol/albuterol hydrofluoroalkane metered dose inhaler (HFA MDI) per day for > 2 consecutive days,
   * exacerbation of asthma.
7. Patients with a history of pneumonectomy or who are planning to undergo thoracotomy for any reason
8. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the six weeks prior to the first screening visit 1
9. Patients with two or more hospitalizations for asthma within the previous twelve months
10. Patients with a recent history of myocardial infarction during the last twelve months or known coronary heart disease that requires treatment
11. Patients with a history of hospitalisation due to heart failure in the past twelve months
12. Patients with myocarditis or any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year
13. Patients with significant alcohol or drug abuse in the opinion of the investigator within the past two years
14. Patients with rheumatoid arthritis or other systemic diseases that require immune system modulating treatment
15. Patients suffering from narrow angle glaucoma with a history of glaucoma, increased intraocular pressure, and/or cataracts
16. Pregnant or nursing women
17. Women of childbearing potential not using a highly effective method of birth control.
18. Patients who have been treated with anti-Immunoglobin-E-antibodies (e.g. omalizumab, Xolair®) or other immune system modulating antibodies such as tumor necrosis factor-alpha blockers within six months prior to Visit 1
19. Patients who have been treated with the following drugs during the past four weeks prior to Visit 1 or are foreseen to need this during the study:

    * Non-selective beta-blockers (topical cardio-selective beta-blocker eye medications for non-narrow angle glaucoma are allowed),
    * Oral or other systemic corticosteroids,
    * Oral beta-agonists,
    * Changes in allergen desensitisation therapy in last 6 months,
    * Immune system modulating agents such as methotrexate or cyclosporine,
    * Inhibitors of cytochrome P450 3A4 such as antifungals (e.g. ketoconazole, itraconazole), antibiotics (e.g. erythromycin) or antiretroviral drugs.
    * Patients who have been treated with leukotriene modifiers, chromones or theophylline within two weeks prior to Visit 1
    * Patients who have been treated with tiotropium within 3 weeks prior to Visit 1

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2011-12-23 (Actual); Study Completion 2011-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (41):
- United States (41):
  - 1248.6.01047 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 1248.6.01023 Boehringer Ingelheim Investigational Site, Fullerton, California
  - 1248.6.01041 Boehringer Ingelheim Investigational Site, Huntington Beach, California
  - 1248.6.01038 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1248.6.01004 Boehringer Ingelheim Investigational Site, Mission Viejo, California
  - 1248.6.01028 Boehringer Ingelheim Investigational Site, Palmdale, California
  - 1248.6.01044 Boehringer Ingelheim Investigational Site, Stockton, California
  - 1248.6.01034 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 1248.6.01015 Boehringer Ingelheim Investigational Site, Centennial, Colorado
  - 1248.6.01035 Boehringer Ingelheim Investigational Site, Aventura, Florida
  - 1248.6.01022 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1248.6.01042 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 1248.6.01051 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 1248.6.01052 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 1248.6.01011 Boehringer Ingelheim Investigational Site, Eagle, Idaho
  - 1248.6.01055 Boehringer Ingelheim Investigational Site, Oak Lawn, Illinois
  - 1248.6.01019 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1248.6.01039 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1248.6.01037 Boehringer Ingelheim Investigational Site, Ypsilanti, Michigan
  - 1248.6.01056 Boehringer Ingelheim Investigational Site, Rolla, Missouri
  - 1248.6.01036 Boehringer Ingelheim Investigational Site, Warrensburg, Missouri
  - 1248.6.01020 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1248.6.01049 Boehringer Ingelheim Investigational Site, Berlin, New Jersey
  - 1248.6.01054 Boehringer Ingelheim Investigational Site, Trenton, New Jersey
  - 1248.6.01010 Boehringer Ingelheim Investigational Site, Verona, New Jersey
  - 1248.6.01006 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1248.6.01031 Boehringer Ingelheim Investigational Site, High Point, North Carolina
  - 1248.6.01045 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1248.6.01005 Boehringer Ingelheim Investigational Site, Gresham, Oregon
  - 1248.6.01021 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1248.6.01013 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1248.6.01040 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1248.6.01012 Boehringer Ingelheim Investigational Site, Upland, Pennsylvania
  - 1248.6.01048 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1248.6.01050 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1248.6.01002 Boehringer Ingelheim Investigational Site, Live Oak, Texas
  - 1248.6.01046 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1248.6.01001 Boehringer Ingelheim Investigational Site, Waco, Texas
  - 1248.6.01025 Boehringer Ingelheim Investigational Site, Murray, Utah
  - 1248.6.01053 Boehringer Ingelheim Investigational Site, Alexandria, Virginia
  - 1248.6.01030 Boehringer Ingelheim Investigational Site, Tacoma, Washington

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, double-blind, double-dummy, Placebo, parallel group study to assess and compare efficacy and safety on an 8-week Treatment with BI 54903 administered via Respimat® inhaler and fluticasone propionate Hydrofluoralkane Metered dose inhaler in patients with asthma.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Oral inhalation from Hydrofluoralkane (HFA) Metered dose inhaler (MDI) (combined with placebo Respimat® inhaler).
- BI 54903 45.5µg Bid: 2 puffs of 22.7 microgram (µg) (total 45.5 µg) of BI 54903 ethanolic solution for inhalation were inhaled orally twice daily (bid), in the morning and evening via Respimat® inhaler (combined with 2 puffs placebo Hydrofluoralkane (HFA) Metered dose inhaler (MDI) bid) for a treatment period of 8 weeks.
- BI 54903 90.9 µg Bid: 2 puffs of 45.5 microgram (µg) (total 90.9 µg) of BI 54903 ethanolic solution for inhalation were inhaled orally twice daily (bid), in the morning and evening via Respimat® inhaler (combined with 2 puffs placebo Hydrofluoralkane (HFA) Metered dose inhaler (MDI) bid) for a treatment period of 8 weeks.
- BI 54903 181.8 µg Bid: 2 puffs of 90.9 microgram (µg) (total 181.8 µg) of BI 54903 ethanolic solution for inhalation were inhaled orally twice daily (bid), in the morning and evening via Respimat® inhaler (combined with 2 puffs placebo Hydrofluoralkane (HFA) Metered dose inhaler (MDI) bid) for a treatment period of 8 weeks.
- Fluticasone Propionate 220µg Bid: 2 puffs of 110 µg (total 220 µg) Fluticasone propionate were orally administered twice daily (bid) via Hydrofluoralkane (HFA) Metered dose inhaler (MDI), combined with placebo Respimat® inhaler.
Period: Overall Study
Arm/Group | Placebo | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid
Started | 6 | 6 | 6 | 7 | 5
Treated | 6 | 6 | 5 | 7 | 5
Completed | 1 | 0 | 0 | 2 | 1
Not Completed | 5 | 6 | 6 | 5 | 4
Not completed — Not treated | 0 | 0 | 1 | 0 | 0
Not completed — Not yet defined | 3 | 6 | 5 | 5 | 4
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were randomised and treated with at least dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 7 | 5 | 6 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (16.4) | 48.4 (6.7) | 53.7 (7.8) | 42.6 (18.2) | 47.8 (8.8) | 47.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 4 | 5 | 15
  Male | 5 | 2 | 5 | 1 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 5 | 4 | 7 | 5 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2 | 1 | 5
  White | 5 | 3 | 7 | 3 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Randomisation Baseline to the End of the 8-week Treatment Period in Trough (Pre-dose and Pre-rescue Bronchodilator) Forced Expiratory Volume in One Second (FEV1)
Description: Mean change from randomisation baseline to the end of the 8-week treatment period in trough (pre-dose and pre-rescue bronchodilator) forced expiratory volume in one second (FEV1).
Time Frame: At baseline and at week 8.
Population: Study was terminated by the decision of sponsor. No valid data for primary and secondary endpoints were collected and no analyses of primary and secondary endpoints were conducted.
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Mean Changes From Randomisation Baseline in Trough (Pre-dose and Pre-rescue Bronchodilator) Forced Vital Capacity (FVC) After 2, 4 and 8-week Treatment Periods
Description: Mean changes from randomisation baseline in trough (pre-dose and pre-rescue bronchodilator) forced vital capacity (FVC) after 2, 4 and 8-week treatment periods.
Time Frame: At baseline and at week 2, 4 and 8.
Population: as for outcome 1
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean Changes From Randomisation Baseline in Trough (Pre-dose and Pre-rescue Bronchodilator) Forced Expiratory Volume in One Second (FEV1) After 2 and 4-week Treatment Periods
Description: Mean changes from randomisation baseline in trough (pre-dose and pre-rescue bronchodilator) forced expiratory volume in one second (FEV1) after 2 and 4-week treatment periods.
Time Frame: At baseline and at week 2 and 4.
Population: as for outcome 1
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Mean Changes From Randomisation Baseline in Trough (Morning Pre-dose and Pre-rescue Bronchodilator) FEF25-75 After 2, 4 and 8-week Treatment Periods
Description: Mean change from randomization baseline in through (morning pre-dose and pre-rescue bronchodilator) Forced expiratory flow between 25% and 75% of vital capacity (FEF 25-75) after 2, 4 and 8-week treatment periods.
Time Frame: At baseline and at week 2, 4 and 8.
Population: as for outcome 1
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Mean Pre-dose (and Pre-rescue) Peak Expiratory Flow (PEF) as Assessed Via Asthma Monitor (AM2+) in the Morning and Evening, of the Last Week of the 8-week Treatment Period
Description: Mean pre-dose (and pre-rescue) peak expiratory flow (PEF) as assessed via Asthma monitor (AM2+) in the morning and evening, of the last week of the 8-week treatment period.
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Mean Rescue Medication Use (Daytime and Night-time) as Assessed Via Asthma Monitor (AM2+) in the Morning and Evening, of the Last Week of the 8-week Treatment Period
Description: Mean rescue medication use (daytime and night-time) as assessed via asthma monitor (AM2+) in the morning and evening, of the last week of the 8-week treatment period.
Time Frame: At week 8.
Population: as for outcome 1
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Mean Change From Randomisation Baseline in Asthma Control Questionnaire (ACQ-6) Scores at Subsequent Study Visits
Description: The Asthma Control Questionnaire (ACQ) consists of 6 patient self-evaluated questions with each question in 7-point scale. The items are equally weighted and the ACQ score is the mean of 6 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of less than or equal to 0.75 indicate well-controlled asthma, scores between 0.76 and less than 1.5 indicate partly controlled asthma, and a score greater than or equal to 1.5 indicates uncontrolled asthma.
Time Frame: At baseline and at week 2, 4 and 8.
Population: as for outcome 1
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Mean Change From Randomisation Baseline in Asthma Quality of Life Questionnaire (AQLQ(S)+12) Scores at Subsequent Study Visits
Description: AQLQ(S)+12 are well established and validated questionnaires to measure control of asthma symptoms and quality of life, which is a patient-reported self-administered outcome questionnaire containing 32 items. Each item is scored on a 7-point scale (1=maximal impairment, 7=no impairment). The 32 items of the questionnaire are averaged to produce one overall quality of life score ranging from 1 (severely impaired) to 7 (not impaired at all). Higher scores indicate better quality of life.
Time Frame: At baseline and at week 2, 4 and 8.
Population: as for outcome 1
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Time to Withdrawal Due to First Asthma Exacerbation
Description: Time to withdrawal due to first Asthma exacerbation.
Time Frame: At week 8.
Population: as for outcome 1
Arm/Group | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization until 8 weeks at end of trial + 2 weeks of follow-up period, up to 10 weeks.
Description: The treated set consists of all randomized patients where at least one dose of study medication was taken.
Arm/Group | Placebo | BI 54903 45.5µg Bid | BI 54903 90.9 µg Bid | BI 54903 181.8 µg Bid | Fluticasone Propionate 220µg Bid
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 4/6 | 3/6 | 3/5 | 3/7 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | BI 54903 45.5µg Bid (N=6) | BI 54903 90.9 µg Bid (N=5) | BI 54903 181.8 µg Bid (N=7) | Fluticasone Propionate 220µg Bid (N=5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated by the decision of the sponsor. As limited data were collected due to early termination and only limited number of patients completed the 8-week treatment period, no analysis of primary and secondary endpoint were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.